CLINICAL TRIAL: NCT02503982
Title: Valganciclovir Dosing in Pediatric Solid Organ Transplant Recipients - a Prospective Study
Brief Title: Valganciclovir Dosing in Pediatric Solid Organ Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 001-14-RMC
Record Dates: First submitted 2015-07-14; First posted 2015-07-21 (Estimated); Results first posted 2016-06-30 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2016-04

CONDITIONS: Infection in Solid Organ Transplant Recipients
MeSH Terms: interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Solid Organ Transplanted children (Experimental): Intervention: treatment with prophylactic oral valganciclovir with a fixed dose of 17 mg/kg once daily for prophylaxis, and stratified dose reductions for impaired renal function. Max dose was 900 mg.
  Interventions: Drug: prophylactic Valganciclovir

INTERVENTIONS:
Drug: prophylactic Valganciclovir — The common practice dose at Schneider Children's Medical Center dosing guidelines of valganciclovir is 17 mg/kg once daily for prophylaxis, with stratified dose reductions for impaired renal function. Max dose was 900 mg.
  Other Names: Valcyte

SUMMARY:
Valganciclovir is extensively used for cytomegalovirus (CMV) infection treatment and prophylaxis after solid organ transplantation (SOT). VGC dosing is problematic in children. valganciclovir has variable absorption and is renally excreted. Area Under the Curve (AUC) (0-24) of 40-60 mcg∙h/L is a predictive pharmacokinetic parameter of efficacy and safety. Dosing based on manufacturer recommendations is supra-therapeutic in most cases. A few published dosing algorithms result in AUC out of range.

Objective: To prospectively validate a Valganciclovir administration dosing regimen and compare it to other dosing algorithms.

Methods: Children after SOT at Schneider Children's Medical Center, the largest tertiary pediatric center in Israel, were prospectively studied, starting Dec 2014. The dosing regimen was derived from Seattle Children's Hospital guidelines; 14-16 mg/kg/dose. For impaired renal function, stratified dose reduction was used. Blood was withdrawn at steady state: 2, 5 and 10 hours post dosing. Drug level was analyzed by high pressure liquid chromatography (HPLC).

DETAILED DESCRIPTION:
Valganciclovir is a novel drug used extensively as a prophylactic, preemptive and treatment agent for cytomegalovirus (CMV) infection after solid organ transplantation (SOT).

It is the valine ester prodrug of Ganciclovir,has a bioavailability of approximately 60%, which is up to 10-fold higher than oral ganciclovir .

Based on the correlation between the Pharmacokinetic (PK) of VGC and its clinical efficacy found in adult studies, AUC (0-24) of approximately 40-60 mcg∙h/mL has been described as predictive PK parameter of efficacy. Considering the mechanism of action of Valganciclovir , relationships of exposure-efficacy and exposure-safety are expected to be similar in children and adults.

In 2009, a new dosing algorithm incorporating both body surface area (BSA) and renal function was introduced by the manufacturer for infants and young children:

Dose (mg) =7 × BSA × CrCl

Very few studies have evaluated this dosing for infants and young children. In 2010 the FDA published a safety alert confirming the excessively high dosage calculated by the dosing algorithm in children with low body weight, low body surface area, and normal serum creatinine. This type of patient was not routinely observed in the clinical trials used to derive and confirm the pediatric dose.

As the body weight decreases and/or as the Creatinine Clearance (CrCl) increases excessively high doses are calculated. There is unproportional variability of doses calculated by the algorithm for infants and young children with normal renal function.

Doses can reach as high as 4 fold higher than the weight-based common dosing.

Objective:

1. To prospectively validate a dosing regimen of Valganciclovir administration
2. and to compare it to other dosing algorithms.

Methods:

This is a prospective study of all pediatric SOT recipients who were treated with oral valganciclovir. The common practice dose at Schneider Children's Medical Center dosing guidelines of valganciclovir is 17 mg/kg once daily for prophylaxis, with stratified dose reductions for impaired renal function as shown in the table. Max dose was 900 mg.

Measurement of valganciclovir levels After three days of consistent oral dosing to ensure steady-state concentrations, drug levels were measured at 2, 5 and 10 h following administration of the dose, and were analyzed at the pharmacologic laboratory of "Asaf HaRofeh Medical Center" using standard HPLC, with a lower limit of detection of 0.5 mcg/mL and a coefficient of variation of <10%. AUCs were calculated using the trapezoidal method.

ELIGIBILITY:
Inclusion Criteria:

1. children and adolescents 0-18 years old
2. Solid Organ Transplantation admitted after transplantation
3. Treatment with prophylactic Valganciclovir
4. Glomerular Filtration Rate (GFR) >= 60 mL/min/1.73 m2

Exclusion Criteria:

1. Treatment with ganciclovir IV
2. Glomerular Filtration Rate (GFR) < 60 mL/min/1.73 m2
3. Imipenem treatment
4. Cluster organ transplanted -

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liat Ashkenazy-Hofnung, MD, Principal Investigator — Schneider's Children Medical center of Isreal
Locations (1):
- Schneider childrens medical center of Isreal, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peled O, Berkovitch M, Rom E, Bilavsky E, Bernfeld Y, Dorfman L, Pappo A, Ziv-Baran T, Brandriss N, Bar-Haim A, Amir J, Ashkenazi-Hoffnung L. Valganciclovir Dosing for Cytomegalovirus Prophylaxis in Pediatric Solid-organ Transplant Recipients: A Prospective Pharmacokinetic Study. Pediatr Infect Dis J. 2017 Aug;36(8):745-750. doi: 10.1097/INF.0000000000001595. PMID 28383392

RESULTS

PARTICIPANT FLOW:
Recruitment Details: conducted at the Schneider Children's Medical Center (SCMC) from December 2014 to August 2015.
Pre-assignment Details: A prospective pharmacokinetic. age <18 years of age, GFR>60 mL/min/1.73m2, solid-organ transplantation and oral VGC prophylaxis for CMV infection
Groups:
- Solid Organ Transplanted Children: Intervention: treatment with prophylactic oral valganciclovir with a fixed dose of 17 mg/kg once daily for prophylaxis. Max dose was 900 mg.
  prophylactic Valganciclovir: The common practice dose at Schneider Children's Medical Center dosing guidelines of valganciclovir is 17 mg/kg once daily for prophylaxis. Max dose was 900 mg.
Period: Overall Study
Arm/Group | Solid Organ Transplanted Children
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Solid Organ Transplanted Children
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 7.3 [2.2 to 11.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC)
Description: Valganciclovir area under the curve (AUC) calculated with the trapezoidal method using drug levels measured at 2, 5 and 10 h, and extrapolated beyond the 10 hour time point to arrive at a 24-hour curve.
Time Frame: drug levels measured at 2, 5 and 10 h following administration of the dose on day 4 creating a 24 hours curve
Measure: Median (Inter-Quartile Range); unit: mcg∙h/mL
Arm/Group | Solid Organ Transplanted Children
Number analyzed (Participants) | 13
mcg∙h/mL | 21.0 [17.1 to 39.8]

ADVERSE EVENTS:
Arm/Group | Solid Organ Transplanted Children
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Organ Transplanted Children (N=13)
Hematologic toxicity (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes